CLINICAL TRIAL: NCT00309257
Title: Effects of an Intensified Treatment With ACE-inhibitors, Angiotensin II Receptor Antagonists and Statins in Alport Syndrome
Brief Title: Effects of an Intensified Treatment With ACE-I,ATA II and Statins in Alport Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVA01
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2009-10

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; benazepril; Valsartan; Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACE inhibitor, ATA II antagonists and Statins (Experimental)
  Interventions: Drug: ACE I, ATA II and Statins; Drug: Benazepril, Valsartan and Fluvastatin

INTERVENTIONS:
Drug: ACE I, ATA II and Statins
Drug: Benazepril, Valsartan and Fluvastatin — Patients will be given a low dose of Benazepril, 10 mg/die,that, if tolerated, will be up-titrated, after a week,to 20 mg/day.
  Patients will be given Valsartan, 80 mg/die,up-titrated after a week to 160 mg/die. Fluvastatin will be started at 40 mg/die.If tolerated, will up-titrated to 80 mg/die. In case of liver, muscular or renal toxicity, fluvastatin will be back-titrated to 40 mg or withdrawn as deemed appropriate.

SUMMARY:
Alport syndrome (AS) represents a form of progressive hereditary nephritis in which the genetic defect resides in the synthesis of one of several subunits of type IV collagen, the predominant constituent of basement membranes in renal glomeruli. Renal impairment occurs with time and severe renal failure with hypertension and uremia represent the end stage of the disease, even if a high variability in the rate of progression is described.Males are usually affected by a progressive form of the disease. Affected females with X-linked syndrome usually have a good prognosis with a mild renal impairment. The disease is also associated to a sensor neural deafness which can occur in approximately half of the patient affected and usually correlates with renal impairment. No definite treatment exists in order to delay the time of dialysis or a kidney transplant. Many studies showed that Angiotensin converting enzyme (ACE) inhibitors slow glomerular filtration rate (GFR) decline and limit progression to end stage renal disease (ERDS) and dialysis in several chronic nephropathies associated with proteinuria. The combination of ACE-I with Angiotensin II receptor antagonists may reduce proteinuria more effectively than the two drugs alone. Moreover the addition of statins may synergize the antiproteinuric effects of ACE-I and ATAII antagonists in experimental models of chronic renal diseases.

The purpose of this study is to evaluate the effect of a standardized multimodal nephroprotection intervention (Remission Clinic) in Alport patients with renal involvement.

DETAILED DESCRIPTION:
Alport syndrome (AS) represents a form of progressive hereditary nephritis in which the genetic defect resides in the synthesis of one of several subunits of type IV collagen, the predominant constituent of basement membranes in glomeruli, eye, cochlea. From a genetical point of view, the disease is quite heterogeneous, since we have X-linked, autosomal recessive and autosomal dominant variants of the syndrome. In most cases (about 80%) the model of inheritance is X-linked and the affected patients are males. Here the mutation stays on X-chromosome in a gene codifying for alpha-5(IV). In about 15% of patients the inheritance is autosomal recessive, with a severe disease both in males and females. The involved genes here are located on chromosome 2 and codifying respectively for alpha-3(IV) and alpha-4(IV) chains. In a 5% the model of inheritance is autosomal dominant and here the deterioration of renal function usually occurs more slowly.

Clinical manifestations include microscopic hematuria as the first finding, which can also became gross hematuria (episodes during upper respiratory infections) or manifest as intermittent (heterozygous females). Another sign is proteinuria of various degrees. It may be from insignificant, described in heterozygous females, or a progressive proteinuria (recessive or X-linked disease). It is evident from clinical studies of Alport patients that a persistent massive proteinuria, inducing a progressive interstitial fibrosis, indicates a very poor prognosis. The presence of glomerular podocytes has been described in urinary sediments of patients with renal diseases, including AS and recent data suggest that podocyturia could act as a marker for estimating the severity of active glomerular injury and as a predictor of disease progression. Renal impairment occurs with time and severe renal failure with hypertension and uremia represent the end stage of the disease, even if an high variability in the rate of progression is described. The prognosis is variable. Males are usually affected by progressive form of disease. Affected females with X-linked syndrome usually have a good prognosis with a mild renal impairment. Some females evolve in a progressive nephritis. The disease is also associated to a sensorineural deafness which can occur in approximately half of the patient affected and usually correlates with renal impairment. Many studies showed that angiotensin converting enzyme (ACE) inhibitors slow glomerular filtration rate (GFR) decline and limit progression to end stage renal disease (ERDS) and dialysis in several chronic nephropathies. ACE inhibitors delay renal fibrosis both by an hemodynamic mechanism (reduction of the intraglomerular hypertension, glomerular hyperfiltration and associated proteinuria) and a non-hemodynamic mechanism (decrease of angiotensin II, a potent inducer of TGF-β release which is a fibrogenic cytokine).

ACE inhibitors given to COL4A3 knockout mouse (a model for autosomal-recessive AS) during pre-symptomatic disease, markedly delayed the onset of proteinuria, progressive renal damage and uremia. Conversely the same treatment did not improve renal outcome in this mouse model if fibrosis and impairment of renal function was already present. These results are in agreement with the findings that ACE inhibitor have beneficial effects against proteinuria, renal function deterioration and survival in Samoyed dogs, a model for X-linked hereditary nephropathy closely mimicking human AS.

Moreover recent clinical data suggest that even in young patients affected by AS a decrease in proteinuria and a stabilization in renal function result from the use of ACE inhibition.

The combination of ACE-I with ATAII antagonists may reduce proteinuria more effectively than the two drugs alone. Moreover the addition of statins may synergize the antiproteinuric effects of ACE-I and ATAII antagonists in experimental models of chronic renal diseases. Statins given with or without inhibitors of the renin-angiotensin-system have an additive effect on reducing proteinuria also in humans.

The purpose of this study is to evaluate the effects of a multimodel treatment including the integrated use of ACE inhibitors (ACE-I), Angiotensin II antagonists (ATA), non dihydropyridinic calcium channel blockers (CCBS) and statins in AS and renal involvement.

Aims of the study Primary To evaluate the effect of a standardized multimodal nephroprotection intervention (Remission Clinic) on overnight urine albumin excretion rate (UAE) in Alport patients with renal involvement Secondary

1. To evaluate the effect of the above treatment on:

   * regression from macro to micro or normoalbuminuria
   * regression from micro to normoalbuminuria
   * regression from high-normal albuminuria to low-normal albuminuria
   * urinary albumin/creatinine ratio
   * systolic/diastolic blood pressure
   * urinary podocyte excretion
   * albumin-IgG-IgM fractional clearances
2. To assess treatment tolerability

ELIGIBILITY:
Inclusion Criteria:

* age ≥15 years
* Alport disease
* Creatinine clearance >20 ml/min/1.73 mq with variation of less than 30% in the three months prior to study entry
* written informed consent. For patients <18 years old a written informed consent of both parents is needed

Exclusion Criteria:

* treatment with immunosuppressive drugs in the six months preceding the study
* vascular disease of the kidney
* obstructive uropathy, prostatic hypertrophy, incomplete bladder emptying
* transplanted kidney
* clinically relevant electrolyte imbalance (e.g., hyperkaliemia with serum K+ > 5.5 mEq/l)
* any concomitant medication with drugs that may directly affect UAE including ACE-inhibitors, angiotensin II receptor antagonists, non dihydropyridine CCBS, HMGCoA reductase inhibitors in the last one month
* history of hypersensitivity to the study drugs
* impossibility to temporary withdrawn ACE-I or ATA II or statins (heart failure, cardiovascular events over the last three months)
* any clinically relevant condition that may affect study participation and/or study results
* pregnancy, ineffective contraception, breast feeding
* inability to fully understand the purposes/risks of the study and/or to provide a written informed consent

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-01; Primary Completion 2008-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Urinary protein excretion | At baseline and monthly

SECONDARY OUTCOMES:
Blood pressure | At baseline, monthly and when deemed clinically appropriate
Urinary podocyte excretion | At baseline and every six months.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Daina, MD, Principal Investigator — Mario Negri Institute for Phrmacological Research
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy